CLINICAL TRIAL: NCT01986010
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Human Cytomegalovirus Vaccine (V160) in Healthy Adults
Brief Title: Safety, Tolerability, and Immunogenicity of the Human Cytomegalovirus Vaccine (V160) in Healthy Adults (V160-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V160-001
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (17):
- HCMV seropositive (+) V160 Low Dose Intramuscular (IM) (Experimental): Participants seropositive for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Low Dose IM
- HCMV seronegative (-) V160 Low Dose IM (Experimental): Participants seronegative for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Low Dose IM
- HCMV+ V160 Medium Dose IM (Experimental): Participants seropositive for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Medium Dose IM
- HCMV- V160 Medium Dose IM (Experimental): Participants seronegative for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Medium Dose IM
- HCMV+ V160 High Dose IM (Experimental): Participants seropositive for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 High Dose IM
- HCMV- V160 Medium Dose plus MAPA 225 µg IM (Experimental): Participants seronegative for HCMV at Baseline will receive vaccination with V160 plus MAPA adjuvant by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Medium Dose plus Merck Aluminum Phosphate Adjuvant (MAPA) 225 µg /dose IM
- HCMV- V160 High Dose IM (Experimental): Participants seronegative for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 High Dose IM
- HCMV+ V160 High Dose plus MAPA 225 µg IM (Experimental): Participants seropositive for HCMV at Baseline will receive vaccination with V160 plus MAPA adjuvant by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 High Dose plus MAPA 225 µg /dose IM
- HCMV+ V160 Maximum Dose IM (Experimental): Participants seropositive for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Maximum Dose IM
- HCMV- V160 High Dose plus MAPA 225 µg IM (Experimental): Participants seronegative for HCMV at Baseline will receive vaccination with V160 plus MAPA adjuvant by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 High Dose plus MAPA 225 µg /dose IM
- HCMV- V160 Maximum Dose IM (Experimental): Participants seronegative for HCMV at Baseline will receive V160 vaccination by IM injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Maximum Dose IM
- HCMV+ Placebo IM (Placebo Comparator): Participants seropositive for HCMV at Baseline will receive placebo by IM injection on Day 1, Month 1, and Month 6
  Interventions: Other: Placebo IM
- HCMV- Placebo IM (Placebo Comparator): Participants seronegative for HCMV at Baseline will receive placebo by IM injection on Day 1, Month 1, and Month 6
  Interventions: Other: Placebo IM
- HCMV+ V160 Medium Dose Intradermal (ID) (Experimental): Participants seropositive for HCMV at Baseline will receive V160 vaccination by ID injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Medium Dose ID
- HCMV- V160 Medium Dose ID (Experimental): Participants seronegative for HCMV at Baseline will receive V160 vaccination by ID injection on Day 1, Month 1, and Month 6
  Interventions: Biological: V160 Medium Dose ID
- HCMV+ Placebo ID (Placebo Comparator): Participants seropositive for HCMV at Baseline will receive placebo by ID injection on Day 1, Month 1, and Month 6
  Interventions: Other: Placebo ID
- HCMV- Placebo ID (Placebo Comparator): Participants seronegative for HCMV at Baseline will receive placebo by ID injection on Day 1, Month 1, and Month 6
  Interventions: Other: Placebo ID

INTERVENTIONS:
Biological: V160 Low Dose IM — V160 administered as a 0.75 mL intramuscular injection
  Arms: HCMV seronegative (-) V160 Low Dose IM; HCMV seropositive (+) V160 Low Dose Intramuscular (IM)
Biological: V160 Medium Dose IM — V160 administered as a 0.75 mL intramuscular injection
  Arms: HCMV+ V160 Medium Dose IM; HCMV- V160 Medium Dose IM
Biological: V160 High Dose IM — V160 administered as a 0.75 mL intramuscular injection
  Arms: HCMV+ V160 High Dose IM; HCMV- V160 High Dose IM
Biological: V160 Medium Dose plus Merck Aluminum Phosphate Adjuvant (MAPA) 225 µg /dose IM — V160 plus MAPA administered as a 0.75 mL intramuscular injection
  Arms: HCMV- V160 Medium Dose plus MAPA 225 µg IM
Biological: V160 High Dose plus MAPA 225 µg /dose IM — V160 plus MAPA administered as a 0.75 mL intramuscular injection
  Arms: HCMV+ V160 High Dose plus MAPA 225 µg IM; HCMV- V160 High Dose plus MAPA 225 µg IM
Biological: V160 Maximum Dose IM — V160 administered as a 0.75 mL intramuscular injection
  Arms: HCMV+ V160 Maximum Dose IM; HCMV- V160 Maximum Dose IM
Other: Placebo IM — Placebo administered as a 0.75 mL intramuscular injection
  Arms: HCMV+ Placebo IM; HCMV- Placebo IM
Biological: V160 Medium Dose ID — V160 administered as a 0.1 mL intradermal injection
  Arms: HCMV+ V160 Medium Dose Intradermal (ID); HCMV- V160 Medium Dose ID
Other: Placebo ID — Placebo administered as a 0.1 mL intradermal injection
  Arms: HCMV+ Placebo ID; HCMV- Placebo ID

SUMMARY:
This study will evaluate the safety, tolerability, and immunogenicity of various doses, formulations, and routes of administration of Human Cytomegalovirus (HCMV) vaccine V160 administered in a 3-dose regimen in healthy adults. The initial treatment arm of HCMV seropositive participants will receive V160 Low Dose without adjuvant by intramuscular injection. Escalation of the V160 dose, inclusion of adjuvant, administration by intradermal injection, and vaccination of HCMV seronegative participants will be performed only after review of safety data of previous treatment arms. The purpose of the study is to identify vaccine formulations associated with optimal safety profile and HCMV-specific immune response for evaluation in subsequent clinical studies of V160.

ELIGIBILITY:
Inclusion Criteria:

* Healthy based on medical history and physical examination
* Serologically confirmed to be HCMV seronegative or HCMV seropositive
* Agrees to avoid unusual, unaccustomed strenuous, vigorous physical exercise/activity from 72 hours before through 72 hours after each dose of study vaccine
* Body weight ≥110 lbs (50 kg) and body mass index (BMI) of 19 to 32 kg/m^2
* If of reproductive potential, agrees to the following during the study and for 4 weeks after the last dose of study vaccine: 1) practice abstinence from heterosexual activity, or 2) use or have their partner use 2 allowable methods of birth control during heterosexual activity

Exclusion Criteria:

* Has previously received any cytomegalovirus vaccine
* Has history of allergic reaction or anaphylactic reaction to any vaccine component that required medical intervention
* Has history of any severe allergic reaction that required medical intervention
* Is pregnant or breastfeeding or expecting to conceive from 2 weeks before the study through 1 month after the last dose of study vaccine
* Plans to donate eggs or sperm from study start through 1 month after the last dose of study drug
* Has impairment of immunologic function including, but not limited to autoimmune disease, splenectomy, or human immunodeficiency virus acquired immunodeficiency syndrome (HIV/AIDS)
* Received systemic corticosteroids for ≥14 consecutive days and has not completed treatment within 30 days of study start
* Received immunosuppressive therapy including, but not limited to rapamycin and equivalents, tacrolimus, FK-506, fujimycin, or other therapies used for solid organ/cell transplant, radiation therapy, immunosuppressive/cytotoxic chemotherapy, or other therapy known to interfere with the immune response within 1 year of study start
* Has a condition in which repeated venipuncture or injections pose more than minimal risk, such as hemophilia, thrombocytopenia or other severe coagulation disorders, or significantly impaired venous access
* Has a condition that requires active medical intervention or monitoring such as diabetes mellitus, autoimmune disease, or a clinically significant chronic medical condition that is considered progressive
* Has history within the past 5 years or current drug or alcohol abuse
* Has major psychiatric illness
* Is legally or mentally incapacitated
* Has participated in another clinical study in the past 4 weeks, or plans during the present study to participate in a treatment-based study or a study in which an invasive procedure is performed
* Has received valganciclovir, ganciclovir, valacyclovir, foscarnet, or cidofovir from 4 weeks prior to 1 month following each V160 vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2016-04-19 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Cox KS, Zhang L, Freed DC, Tang A, Zhang S, Zhou Y, Wang IM, Rupp RE, Adler SP, Musey LK, Wang D, Vora KA, Fu TM. Functional Evaluation and Genetic Evolution of Human T-Cell Responses After Vaccination With a Conditionally Replication-Defective Cytomegalovirus Vaccine. J Infect Dis. 2021 Jun 4;223(11):2001-2012. doi: 10.1093/infdis/jiaa631. PMID 33031517
- [Derived] Adler SP, Lewis N, Conlon A, Christiansen MP, Al-Ibrahim M, Rupp R, Fu TM, Bautista O, Tang H, Wang D, Fisher A, Culp T, Das R, Beck K, Tamms G, Musey L; V160-001 Study Group. Phase 1 Clinical Trial of a Conditionally Replication-Defective Human Cytomegalovirus (CMV) Vaccine in CMV-Seronegative Subjects. J Infect Dis. 2019 Jul 2;220(3):411-419. doi: 10.1093/infdis/jiz141. PMID 31535143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy males and females age 18 years of age and older were enrolled in this trial.
Groups:
- HCMV Seropositive (+) V160 10u Intramuscular (IM): Participants seropositive for Human cytomegalovirus (HCMV) at Baseline received 10 units (u) V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV + V160 30u IM: Participants seropositive for HCMV at Baseline received 30u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV+ V160 100u IM: Participants seropositive for HCMV at Baseline received 100u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV+ V160 100u MAPA IM: Participants seropositive for HCMV at Baseline received 100u V160 plus Merck Aluminum Phosphate Adjuvant (MAPA) adjuvant vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV+ V160 250u IM: Participants seropositive for HCMV at Baseline received 250u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV+ Placebo IM: Participants seropositive for HCMV at Baseline received placebo vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV+ V160 30u ID: Participants seropositive for HCMV at Baseline received 30u V160 vaccination by intradermal (ID) injection on Day 1, Month 1, and Month 6
- HCMV+ Placebo ID: Participants seropositive for HCMV at Baseline received vaccination with placebo by ID injection on Day 1, Month 1, and Month 6
- HCMV Seronegative (-) V160 10u IM: Participants seronegative for HCMV at Baseline received 10u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 30u IM: Participants seronegative for HCMV at Baseline received vaccination with 30u V160 by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 30u MAPA IM: Participants seronegative for HCMV at Baseline received 30u V160 plus MAPA adjuvant vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 100u IM: Participants seronegative for HCMV at Baseline received 100u V160 by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 100u MAPA IM: Participants seronegative for HCMV at Baseline received 100u V160 plus MAPA adjuvant by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 250u IM: Participants seronegative for HCMV at Baseline received 250u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 Placebo IM: Participants seronegative for HCMV at Baseline received placebo vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 30u ID: Participants seronegative for HCMV at Baseline received 30u V160 by ID injection on Day 1, Month 1, and Month 6
- HCMV- Placebo ID: Participants seronegative for HCMV at Baseline received placebo by ID injection on Day 1, Month 1, and Month 6
Period: Overall Study
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Started | 13 | 14 | 14 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Vaccination 1 | 13 | 14 | 14 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Vaccination 2 | 12 | 13 | 12 | 10 | 9 | 19 | 10 | 4 | 11 | 10 | 10 | 10 | 10 | 9 | 16 | 10 | 4
Vaccination 3 | 10 | 10 | 9 | 10 | 9 | 15 | 10 | 4 | 10 | 10 | 10 | 8 | 10 | 9 | 13 | 10 | 4
Completed | 7 | 6 | 7 | 8 | 6 | 11 | 10 | 4 | 6 | 7 | 3 | 1 | 0 | 0 | 6 | 0 | 0
Not Completed | 6 | 8 | 7 | 2 | 5 | 8 | 0 | 0 | 6 | 3 | 7 | 10 | 10 | 11 | 10 | 11 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2 | 2 | 2 | 0 | 0 | 4 | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Not completed — Status Not Recorded | 2 | 4 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 7 | 7 | 9 | 9 | 5 | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- HCMV Seropositive (+) V160 10u Intramuscular (IM): Participants seropositive for Human cytomegalovirus (HCMV) at Baseline received 10u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- Total: Total of all reporting groups
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID | Total
Number analyzed (Participants) | 13 | 14 | 14 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (14.8) | 47.7 (14.5) | 44.9 (13.2) | 48.8 (10.6) | 46.4 (13.7) | 46.5 (15.1) | 51.7 (18.9) | 47.5 (16.7) | 45.0 (11.8) | 32.5 (10.9) | 39.0 (16.6) | 41.1 (14.5) | 53.1 (10.7) | 40.0 (14.4) | 44.9 (15.7) | 36.1 (12.7) | 31.5 (13.1) | 44.1 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 9 | 6 | 7 | 10 | 6 | 2 | 7 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 2 | 109
  Male | 6 | 5 | 5 | 4 | 4 | 9 | 4 | 2 | 5 | 4 | 4 | 5 | 4 | 5 | 8 | 5 | 2 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 2 | 1 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 19
  Not Hispanic or Latino | 9 | 13 | 12 | 8 | 10 | 19 | 7 | 4 | 10 | 10 | 8 | 11 | 10 | 9 | 15 | 11 | 4 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 3 | 6 | 4 | 5 | 8 | 0 | 1 | 3 | 2 | 2 | 1 | 1 | 2 | 4 | 1 | 0 | 47
  White | 7 | 10 | 7 | 6 | 5 | 8 | 9 | 3 | 8 | 7 | 7 | 10 | 8 | 9 | 10 | 10 | 3 | 127
  More than one race | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 2 weeks after vaccination on Day 1, Month 1 and Month 6 (up to Day 15, Week 6 and Week 26)
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 75.0 | 92.9 | 84.6 | 100.0 | 100.0 | 57.9 | 100.0 | 50.0 | 75.0 | 90.0 | 90.0 | 100.0 | 90.0 | 90.9 | 56.3 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants With an Injection-site AE
Description: Injection-site AEs are defined as redness, swelling, and pain/tenderness.
Time Frame: Up to 2 weeks after vaccination on Day 1, Month 1 and Month 6 (up to Day 15, Week 6 and Week 26)
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 58.3 | 85.7 | 69.2 | 80.0 | 100.0 | 26.3 | 90.0 | 0.0 | 66.7 | 80.0 | 80.0 | 90.9 | 90.0 | 81.8 | 31.3 | 100.0 | 50.0

3. Primary Outcome: Percentage of Participants With a Systemic AE
Description: A Systemic AE includes, but is not exclusive of, the following AEs: fatigue, myalgia, headache and joint pain
Time Frame: Up to 2 weeks after vaccination on Day 1, Month 1 and Month 6 (up to Day 15, Week 6 and Week 26)
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 66.7 | 64.3 | 69.2 | 90.0 | 90.9 | 57.9 | 80.0 | 50.0 | 66.7 | 90.0 | 70.0 | 100.0 | 70.0 | 90.9 | 56.3 | 100.0 | 100.0

4. Primary Outcome: Percentage of Participants With a Serious Adverse Event (SAE)
Description: A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event
Time Frame: Up to 2 weeks after vaccination on Day 1, Month 1 and Month 6 (up to Day 15, Week 6 and Week 26)
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With a Serious Vaccine-Related Adverse Event
Description: A serious adverse event is any adverse event occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. A serious vaccine-related adverse event was determined by the investigator to be related to the vaccine.
Time Frame: Up to 2 weeks after vaccination on Day 1, Month 1 and Month 6 (up to Day 15, Week 6 and Week 26)
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Month 6
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9.1 | 0 | 9.1 | 0 | 9.1 | 0

7. Primary Outcome: Percentage of Participants With Events of Clinical Interest (ECI)
Description: An event of clinical interest (ECI) is identified as any overdose, elevated liver values meeting threshold criteria (aspartate aminotransferase or alanine aminotransferase ≥3x upper limit of normal (ULN); total bilirubin ≥2x ULN, and, at the same time, alkaline phosphatase <2xULN). Additionally, confirmed, diagnosed autoimmune conditions are considered ECIs.
Time Frame: Up to 18 months
Population: All randomized participants who received at least 1 vaccination and had follow-up safety data available
Measure: Number; unit: Percentage of participants
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ Placebo IM | HCMV+ V160 30u ID | HCMV+ Placebo ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- Placebo ID
Number analyzed (Participants) | 12 | 14 | 13 | 10 | 11 | 19 | 10 | 4 | 12 | 10 | 10 | 11 | 10 | 11 | 16 | 11 | 4
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Geometric Mean Titer of HCMV-specific Neutralizing Antibody After Vaccination 3
Description: Serum samples for measuring neutralizing antibodies using the Merck Neutralizing Antibody (NAb) assay were collected at month 7. The LiCor-based near-infrared dye (NIRDye) In-Cell Western (ICW) HCMV microneutralization assay was used to detect and quantify anti-HCMV neutralizing antibodies. The primary hypothesis was that for HCMV-seronegative participants, at least 1 of the vaccination groups receiving V160 formulated with or without adjuvant would exhibit higher HCMV-specific neutralizing antibody titers than the placebo group.
Time Frame: Month 7 (1 month after vaccination 3 at Month 6)
Population: All randomized participants who received at least 1 dose of the study vaccine or placebo and had at least 1 valid neutralizing antibody result.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Groups:
- HCMV+ Placebo IM or ID: Participants seropositive for HCMV at Baseline received vaccination with placebo by IM or ID injection on Day 1, Month 1, and Month 6
- HCMV- Placebo IM or ID: Participants seronegative for HCMV at Baseline received placebo by IM or ID injection on Day 1, Month 1, and Month 6
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ V160 30u ID | HCMV+ Placebo IM or ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 30u ID | HCMV- Placebo IM or ID
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 9 | 9 | 19 | 10 | 10 | 10 | 9 | 9 | 10 | 11 | 19
Geometric Mean Titer | 3301 [2097 to 5197] | 4177 [2721 to 6412] | 7740 [4190 to 14297] | 5701 [3526 to 9218] | 3535 [2115 to 5907] | 8601 [5305 to 13944] | 2224 [1522 to 3249] | 328 [210 to 511] | 1532 [1075 to 2182] | 1361 [886 to 2090] | 820 [524 to 1285] | 2573 [1863 to 3553] | 1241 [699 to 2203] | 1261 [733 to 2169] | 20 [20 to 20]
Statistical Analysis 1: Comparison: HCMV Seropositive (+) V160 10u Intramuscular (IM) vs HCMV+ Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; GMT Ratio = 1.5, 95% CI 2-sided [0.8 to 2.6]
Statistical Analysis 2: Comparison: HCMV + V160 30u IM vs HCMV+ Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; GMT Ratio = 1.9, 95% CI 2-sided [1.1 to 3.2]
Statistical Analysis 3: Comparison: HCMV+ V160 100u IM vs HCMV+ Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; GMT Ratio = 3.5, 95% CI 2-sided [1.6 to 7.4]
Statistical Analysis 4: Comparison: HCMV+ V160 100u MAPA IM vs HCMV+ Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; GMT Ratio = 2.6, 95% CI 2-sided [1.4 to 4.6]
Statistical Analysis 5: Comparison: HCMV+ V160 250u IM vs HCMV+ Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; GMT Ratio = 1.6, 95% CI 2-sided [0.9 to 3.0]
Statistical Analysis 6: Comparison: HCMV+ V160 30u ID vs HCMV+ Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; GMT Ratio = 3.9, 95% CI 2-sided [2.2 to 7.0]
Statistical Analysis 7: Comparison: HCMV Seronegative (-) V160 10u IM vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 16.4, 95% CI 2-sided [9.5 to 28.4]
Statistical Analysis 8: Comparison: HCMV- V160 30u IM vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 76.6, 95% CI 2-sided [49.5 to 118.6]
Statistical Analysis 9: Comparison: HCMV- V160 30u MAPA IM vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 68.1, 95% CI 2-sided [40.1 to 115.6]
Statistical Analysis 10: Comparison: HCMV- V160 100u IM vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 41.0, 95% CI 2-sided [23.8 to 70.7]
Statistical Analysis 11: Comparison: HCMV- V160 100u MAPA IM vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 128.6, 95% CI 2-sided [87.0 to 190.3]
Statistical Analysis 12: Comparison: HCMV- V160 250u IM vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 62.0, 95% CI 2-sided [30.5 to 126.1]
Statistical Analysis 13: Comparison: HCMV- V160 30u ID vs HCMV- Placebo IM or ID; GMT Ratio: GMT V160/GMT placebo; Test type: Other; p < 0.001, Two sample t-test — Hypothesis is GMT Ratio >1; GMT Ratio = 63.0, 95% CI 2-sided [31.9 to 124.6]

9. Secondary Outcome: Geometric Mean Count of Peripheral Blood Mononuclear Cells Secreting Interferon-Gamma
Description: In order to evaluate the cellular immune response to the vaccine(s), the HCMV enzyme-linked immunospot (ELISPOT) assay was used to detect interferon gamma (IFN-γ) secreting HCMV-specific cells from peripheral blood mononuclear cells (PBMCs). Results are expressed as the frequency of spot forming cells (SFCs) per million PBMCs (SFC/10^6 PBMCs). Results are presented for the following HCMV proteins: pp65, Immediate early Protein 1 (IE1), Immediate early Protein 2 (IE2), Glycoprotein B (gB), and also for purified HCMV virion stock.
Time Frame: Month 7 (1 month after vaccination 3 at Month 6)
Population: All randomized participants who received at least 1 dose of the study vaccine or placebo and had at least 1 valid PBMC interferon-gamma result.
Measure: Geometric Mean (95% Confidence Interval); unit: SFC/10^6 PBMCs
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ V160 30u ID | HCMV+ Placebo IM or ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 30u ID | HCMV- Placebo IM or ID
Number analyzed (Participants) | 9 | 10 | 10 | 6 | 8 | 10 | 18 | 8 | 7 | 10 | 6 | 8 | 10 | 7 | 17
SFC/10^6 PBMCs
  pp65 | 819 [362 to 1853] | 419 [174 to 1007] | 1384 [66 to 2873] | 1105 [422 to 2892] | 1206 [565 to 2573] | 1080 [570 to 2047] | 800 [457 to 1401] | 886 [394 to 1993] | 468 [195 to 1125] | 865 [429 to 1745] | 380 [144 to 999] | 1325 [656 to 2679] | 512 [174 to 1502] | 1145 [530 to 2474] | 19 [11 to 34]
  IE1 | 855 [262 to 2786] | 340 [85 to 1353] | 419 [106 to 1660] | 370 [79 to 1719] | 417 [116 to 1507] | 379 [111 to 1299] | 200 [75 to 533] | 776 [310 to 1943] | 358 [123 to 1043] | 913 [416 to 2003] | 577 [158 to 2099] | 933 [384 to 2264] | 742 [326 to 1688] | 1796 [702 to 4590] | 12 [6 to 24]
  IE2: number analyzed (Participants) | 9 | 10 | 8 | 6 | 8 | 10 | 18 | 8 | 7 | 10 | 5 | 8 | 9 | 7 | 17
  IE2 | 122 [48 to 312] | 101 [47 to 216] | 309 [151 to 631] | 72 [34 to 156] | 93 [32 to 271] | 32 [18 to 55] | 49 [32 to 74] | 119 [45 to 313] | 22 [8 to 62] | 34 [15 to 80] | 146 [35 to 609] | 86 [32 to 228] | 131 [52 to 330] | 194 [66 to 576] | 10 [4 to 22]
  gB: number analyzed (Participants) | 9 | 10 | 8 | 6 | 8 | 10 | 18 | 8 | 7 | 10 | 6 | 8 | 9 | 7 | 17
  gB | 195 [69 to 555] | 287 [74 to 1117] | 1137 [422 to 3063] | 217 [58 to 806] | 253 [84 to 761] | 294 [101 to 852] | 140 [64 to 306] | 105 [58 to 190] | 14 [6 to 32] | 38 [22 to 66] | 185 [73 to 469] | 86 [45 to 165] | 135 [73 to 249] | 174 [89 to 339] | 18 [11 to 29]
  Virus: number analyzed (Participants) | 9 | 10 | 9 | 6 | 8 | 10 | 18 | 8 | 7 | 10 | 6 | 8 | 10 | 7 | 17
  Virus | 1190 [544 to 2605] | 384 [114 to 1294] | 2134 [995 to 4578] | 1348 [481 to 3772] | 1708 [732 to 3988] | 937 [430 to 2044] | 1357 [714 to 2579] | 668 [334 to 1334] | 79 [28 to 224] | 268 [135 to 534] | 621 [276 to 1400] | 777 [420 to 1439] | 413 [150 to 1139] | 1160 [597 to 2253] | 17 [10 to 27]

10. Secondary Outcome: Geometric Mean Concentration of Interferon-Gamma After Stimulation of Whole Blood Sample With Pooled HCMV Antigen Peptides
Description: In response to HCMV-specific stimulation of whole blood specimens the whole Blood Cytokine Stimulation (WBStim) assay was used to detect the secretion of interferon gamma (IFN -γ) by an ELISA assay. Results are presented for the following HCMV proteins: pp65, IE1, and gB.
Time Frame: Month 7 (1 month after vaccination 3 at Month 6)
Population: All randomized participants who received at least 1 dose of the study vaccine or placebo and had at least 1 valid whole blood interferon-gamma result.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ V160 30u ID | HCMV+ Placebo IM or ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 30u ID | HCMV- Placebo IM or ID
Number analyzed (Participants) | 10 | 7 | 6 | 7 | 6 | 9 | 15 | 8 | 8 | 9 | 9 | 6 | 7 | 7 | 13
ug/mL
  pp65: number analyzed (Participants) | 10 | 7 | 6 | 7 | 6 | 9 | 14 | 8 | 8 | 8 | 9 | 6 | 7 | 7 | 13
  pp65 | 168 [63 to 445] | 193 [65 to 571] | 79 [26 to 242] | 86 [35 to 209] | 211 [90 to 492] | 64 [30 to 136] | 112 [60 to 210] | 64 [33 to 122] | 97 [53 to 176] | 24 [11 to 56] | 89 [51 to 156] | 8 [5 to 14] | 28 [14 to 56] | 24 [14 to 39] | 5 [3 to 7]
  IE1 | 90 [21 to 389] | 70 [14 to 364] | 13 [2 to 74] | 35 [6 to 217] | 20 [4 to 109] | 27 [7 to 104] | 24 [7 to 82] | 62 [26 to 148] | 35 [20 to 62] | 28 [14 to 55] | 40 [17 to 96] | 11 [5 to 23] | 45 [20 to 101] | 40 [22 to 72] | 5 [3 to 8]
  gB: number analyzed (Participants) | 10 | 6 | 5 | 5 | 6 | 9 | 15 | 7 | 7 | 9 | 9 | 5 | 7 | 5 | 12
  gB | 53 [16 to 175] | 40 [8 to 202] | 64 [11 to 375] | 27 [3 to 213] | 27 [6 to 115] | 62 [18 to 214] | 16 [6 to 48] | 7 [4 to 11] | 10 [6 to 19] | 5 [3 to 9] | 7 [4 to 12] | 10 [6 to 16] | 9 [6 to 16] | 5 [3 to 9] | 6 [4 to 8]

11. Secondary Outcome: Geometric Mean Titer of HCMV-specific Neutralizing Antibody After Vaccinations 1 and 2
Description: Serum samples for measuring neutralizing antibodies using the Merck NAb assay were collected at months 1 and 2. The LiCor-based near-infrared dye (NIRDye) In-Cell Western (ICW) HCMV microneutralization assay was used to detect and quantify anti-HCMV neutralizing antibodies. Values below the lower limit of titer are represented by NA.
Time Frame: Month 1 and 2 (one month after vaccination 1 [Day 1] and vaccination 2 [Month 1])
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | HCMV Seropositive (+) V160 10u Intramuscular (IM) | HCMV + V160 30u IM | HCMV+ V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV+ V160 250u IM | HCMV+ V160 30u ID | HCMV+ Placebo IM or ID | HCMV Seronegative (-) V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 30u ID | HCMV- Placebo IM or ID
Number analyzed (Participants) | 12 | 14 | 12 | 10 | 9 | 10 | 23 | 11 | 10 | 10 | 11 | 10 | 10 | 10 | 20
Geometric Mean Titer
  Month 1 | 3124 [1887 to 5172] | 5186 [3252 to 8270] | 6232 [3764 to 10318] | 6695 [3854 to 11631] | 3831 [2140 to 6858] | 9127 [5253 to 15855] | 2335 [1485 to 3671] | 73 [NA to 137] — Values below the lower limit of titer are represented by NA. | 95 [50 to 184] | 65 [NA to 125] — Values below the lower limit of titer are represented by NA. | 91 [49 to 170] | 134 [70 to 258] | 281 [146 to 542] | 183 [95 to 351] | NA [NA to NA] — Values below the lower limit of titer are represented by NA.
  Month 2: number analyzed (Participants) | 11 | 14 | 10 | 10 | 9 | 10 | 22 | 11 | 10 | 10 | 11 | 10 | 10 | 10 | 20
  Month 2 | 3144 [1893 to 5221] | 5443 [3472 to 8533] | 6959 [4088 to 11845] | 7022 [4126 to 11953] | 4261 [2432 to 7464] | 9412 [5529 to 16021] | 2313 [1468 to 3644] | 143 [89 to 230] | 264 [160 to 433] | 264 [161 to 433] | 288 [180 to 463] | 590 [359 to 968] | 589 [359 to 968] | 451 [275 to 741] | NA [NA to NA] — Values below the lower limit of titer are represented by NA.

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: All randomized participants who received at least 1 vaccination
Groups:
- HCMV + V160 10u IM: Participants seropositive for HCMV at Baseline received 10u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV + V160 100u IM: Participants seropositive for HCMV at Baseline received 100u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV+ V160 100u MAPA IM: Participants seropositive for HCMV at Baseline received 100u V160 plus MAPA adjuvant vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV + V160 250u IM: Participants seropositive for HCMV at Baseline received 250u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV + V160 30u ID: Participants seropositive for HCMV at Baseline received 30u V160 vaccination by ID injection on Day 1, Month 1, and Month 6
- HCMV+ Placebo ID: Participants seropositive for HCMV at Baseline received placebo vaccination by ID injection on Day 1, Month 1, and Month 6
- HCMV- V160 10u IM: Participants seronegative for HCMV at Baseline received 10u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 30u IM: Participants seronegative for HCMV at Baseline received 30u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 100u IM: Participants seronegative for HCMV at Baseline received 100u V160 vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 100u MAPA IM: Participants seronegative for HCMV at Baseline received 100u V160 plus MAPA adjuvant vaccination by IM injection on Day 1, Month 1, and Month 6
- HCMV- V160 30u ID: Participants seronegative for HCMV at Baseline received 30u V160 vaccination by ID injection on Day 1, Month 1, and Month 6
- HCMV- V160 Placebo ID: Participants seronegative for HCMV at Baseline received placebo vaccination by ID injection on Day 1, Month 1, and Month 6
Arm/Group | HCMV + V160 10u IM | HCMV + V160 30u IM | HCMV + V160 100u IM | HCMV+ V160 100u MAPA IM | HCMV + V160 250u IM | HCMV+ Placebo IM | HCMV + V160 30u ID | HCMV+ Placebo ID | HCMV- V160 10u IM | HCMV- V160 30u IM | HCMV- V160 30u MAPA IM | HCMV- V160 100u IM | HCMV- V160 100u MAPA IM | HCMV- V160 250u IM | HCMV- V160 Placebo IM | HCMV- V160 30u ID | HCMV- V160 Placebo ID
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/14 | 0/10 | 0/11 | 0/19 | 0/10 | 0/4 | 0/12 | 0/10 | 0/10 | 0/11 | 0/10 | 0/11 | 0/16 | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/14 | 0/10 | 0/11 | 0/19 | 0/10 | 0/4 | 0/12 | 0/10 | 0/10 | 0/11 | 0/10 | 0/11 | 0/16 | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 9/13 | 13/14 | 12/14 | 10/10 | 11/11 | 12/19 | 10/10 | 2/4 | 9/12 | 9/10 | 9/10 | 11/11 | 9/10 | 10/11 | 10/16 | 11/11 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCMV + V160 10u IM (N=13) | HCMV + V160 30u IM (N=14) | HCMV + V160 100u IM (N=14) | HCMV+ V160 100u MAPA IM (N=10) | HCMV + V160 250u IM (N=11) | HCMV+ Placebo IM (N=19) | HCMV + V160 30u ID (N=10) | HCMV+ Placebo ID (N=4) | HCMV- V160 10u IM (N=12) | HCMV- V160 30u IM (N=10) | HCMV- V160 30u MAPA IM (N=10) | HCMV- V160 100u IM (N=11) | HCMV- V160 100u MAPA IM (N=10) | HCMV- V160 250u IM (N=11) | HCMV- V160 Placebo IM (N=16) | HCMV- V160 30u ID (N=11) | HCMV- V160 Placebo ID (N=4)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 6 (9) | 9 (13) | 7 (19) | 8 (22) | 8 (19) | 9 (15) | 6 (22) | 1 (1) | 7 (15) | 5 (9) | 5 (13) | 6 (20) | 6 (18) | 10 (37) | 8 (16) | 8 (27) | 2 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 1 (2) | 3 (3) | 2 (2) | 2 (4) | 3 (3) | 9 (26) | 0 (0) | 2 (4) | 1 (3) | 3 (5) | 3 (4) | 3 (3) | 3 (6) | 0 (0) | 11 (32) | 2 (2)
Injection site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site joint pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 6 (13) | 12 (31) | 10 (18) | 7 (21) | 11 (35) | 5 (10) | 7 (16) | 0 (0) | 8 (13) | 8 (28) | 8 (19) | 10 (24) | 8 (28) | 9 (35) | 5 (11) | 9 (23) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 9 (18) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site scab (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (5) | 3 (5) | 1 (1) | 9 (27) | 0 (0) | 3 (5) | 1 (3) | 2 (4) | 3 (5) | 4 (9) | 3 (4) | 1 (1) | 11 (34) | 0 (0)
Injection site ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 4 (4) | 3 (11) | 5 (6) | 2 (2) | 3 (10) | 0 (0) | 5 (7) | 2 (3) | 4 (8) | 5 (5) | 3 (7) | 6 (8) | 3 (4) | 5 (14) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (6) | 6 (8) | 5 (13) | 6 (14) | 5 (6) | 4 (10) | 1 (1) | 5 (9) | 7 (12) | 5 (10) | 9 (18) | 5 (12) | 8 (20) | 4 (5) | 4 (13) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (11) | 4 (4) | 6 (14) | 8 (20) | 6 (9) | 7 (13) | 6 (21) | 0 (0) | 5 (10) | 7 (18) | 4 (13) | 9 (17) | 4 (15) | 8 (20) | 5 (8) | 9 (27) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.